CLINICAL TRIAL: NCT05580848
Title: Wrist Arthroscopy During Surgical Treatment of Distal Radius Fractures Improves Functional Outcome: a Randomized Controlled Trial
Brief Title: Wrist Arthroscopy During Surgical Treatment of Distal Radius Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Clinic for Orthopedics Lovran (Other)
Collaborators: University of Rijeka, The Faculty of Medicine (Unknown)
Responsible Party: Principal Investigator, Borjan Josifovski, Principal Investigator, Clinic for Orthopedics Lovran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ClinicOL
Record Dates: First submitted 2022-10-01; First posted 2022-10-14 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Fracture; Radius Fracture Distal
Keywords: Arthroscopy; Radius Fractures; Surveys and Questionnaires; Treatment Outcome; Wrist
MeSH Terms: conditions — Fractures, Bone; Wrist Fractures; Radius Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Examined group (Experimental): 28 patients with indication for distal radius fracture (DRF) osteosynthesis : 14 patients with extraarticular DRF and 14 patients with intraarticular DRF with associated wrist arthroscopy
  Interventions: Procedure: Wrist arthroscopy
- Control group (No Intervention): 28 patients with indication for distal radius fracture (DRF) osteosynthesis : 14 patients with extraarticular DRF and 14 patients with intraarticular DRF without associated wrist arthroscopy.

INTERVENTIONS:
Procedure: Wrist arthroscopy — Wrist arthroscopy is a minimally invasive endoscopic method that enables the diagnosis and treatment of certain diseases and injuries of the radiocarpal, mediocarpal and distal radioulnar joints.
  Wrist arthroscopy enables a direct view of the articular surface of the wrist and the assessment and adequate treatment of articular fractures The wrist arthroscopy procedure also enables the detection and necessary treatment of associated soft tissue injuries (scapho-lunate and/or luno-triquetral ligament, i.e. triangular fibrocartilaginous complex) and/or cartilage lesions in extra-articular and articular fractures.
  Arms: Examined group

SUMMARY:
Wrist arthroscopy (WA) is a potentially useful adjuvant procedure in the surgical treatment (osteosynthesis) of distal radius fractures (DRFs). Previous research on the contribution of WA to DRF treatment has shown different results.

Objectives of the study: (1) Validate wrist functional outcome questionnaires; (2) To determine whether arthroscopically assisted repositioning of fracture fragments in articular DRFs leads to a better treatment outcome; (3) To determine whether arthroscopic observation and treatment of associated soft tissue and / or cartilage injuries in articular DRFs leads to a better treatment outcome; (4) To determine whether arthroscopic observation and treatment of associated soft tissue and / or cartilage injuries in extraarticular DRFs leads to a better treatment outcome.

Research hypotheses: (1) Validated questionnaires will have satisfactory measurement properties (validity, reliability) and will be able to be used in a WA randomized controlled trial; (2) WA as an adjunct to DRF osteosynthesis improves the clinical outcome of treatment.

Subjects: 56 female patients with indication for DRF osteosynthesis aged 50-69 years divided into 2 groups: 1. examined - 28 patients with indication for DRF osteosynthesis (14 patients with extraarticular DRF and 14 patients with intraarticular DRF) with associated WA, and 2. control - 28 patients with indication for DRF osteosynthesis (14 patients with extraarticular DRF and 14 patients with intraarticular DRF) without associated WA.

Methods: As a primary outcome measure, functional outcomes of treatment will be analyzed with the Disabilities of the Arm, Shoulder and Hand (DASH) Score at 3 and 6 months after surgery. As a secondary outcome measures it will be analyzed pain level according to a visual analog scale (VAS), preoperative and postoperative radiographic parameters of distal radius, and clinical outcomes of treatment with the Mayo Wrist Score (MWS) and Patient-Rated Wrist Evaluation (PRWE) score at 3 and 6 months after surgery. Expected scientific contribution: providing answers on the role of WA in the treatment of DRF and associated injuries as well as its impact on treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Distal radius fractures with an indication for surgical treatment according to the AO/OTA classification of patients aged 50-69 years who have signed an informed consent to participate in the research.

Exclusion Criteria:

* Distal radius fractures( DRF) that have an indication for surgical treatment in all patients and in patients younger than 50 and older than 69,
* DRF that do not have an indication for surgical treatment,
* Refusal to participate in the research,
* Inability to decide independently about participation in the research (persons under guardianship),
* Open fractures,
* Presence of severe soft tissue injuries,
* Infections,
* Poor general condition of patients and internal medicine contraindications.

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-11-20 (Estimated); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
DASH Score | 3 months after surgery
  Disabilities of the Arm, Shoulder and Hand It consists of 30 questions and is used to assess functional disorders of the upper extremity. 21 questions examine the extent to which the patient had problems performing certain activities during the last week. 6 questions assess specific symptoms (eg, pain, paresthesias, sleep disturbances) during the last week, and 3 questions assess social or occupational limitations during the last week. The possible score ranges from 0 to 100 points. 0 points represents complete, unrestricted function of the upper extremities, while 100 points represents the greatest possible functional impairment.
DASH Score | 6 months after surgery
  Disabilities of the Arm, Shoulder and Hand It consists of 30 questions and is used to assess functional disorders of the upper extremity. 21 questions examine the extent to which the patient had problems performing certain activities during the last week. 6 questions assess specific symptoms (eg, pain, paresthesias, sleep disturbances) during the last week, and 3 questions assess social or occupational limitations during the last week. The possible score ranges from 0 to 100 points. 0 points represents complete, unrestricted function of the upper extremities, while 100 points represents the greatest possible functional impairment.

SECONDARY OUTCOMES:
VAS | 3 months after surgery.
  The visual analogue scale (VAS) of pain will be used in this study as a tool to assess the clinical outcome of treatment. It consists of the length of a solid line with values at the beginning and end of the line from 0 to 10 cm (0 - 100 mm). The leftmost side means the absence of pain, and the rightmost side means unbearable pain.
VAS | 6 months after surgery.
  The visual analogue scale (VAS) of pain will be used in this study as a tool to assess the clinical outcome of treatment. It consists of the length of a solid line with values at the beginning and end of the line from 0 to 10 cm (0 - 100 mm). The leftmost side means the absence of pain, and the rightmost side means unbearable pain.
MWS | 3 months after surgery.
  The Mayo Wrist Score (MWS) will be evaluated through 4 questions: (1) pain intensity, (2) functional status - ability to return to regular work, (3) active range of motion of bending /extension of the affected wrist compared to the contralateral side (5 answers offered to be scored from 0 to 25 points) and (4) grip strength of the affected hand compared to the contralateral side (5 answers offered to be scored from 0 to 25 points). The possible score ranges from 0 to 100 points. Interpretation of the results: from 90-100 points is an excellent result, 80-90 points is a good result, 60-80 points is a satisfactory result, and below 60 points is a bad result.
MWS | 6 months after surgery.
  The Mayo Wrist Score (MWS) will be evaluated through 4 questions: (1) pain intensity, (2) functional status - ability to return to regular work, (3) active range of motion of bending /extension of the affected wrist compared to the contralateral side (5 answers offered to be scored from 0 to 25 points) and (4) grip strength of the affected hand compared to the contralateral side (5 answers offered to be scored from 0 to 25 points). The possible score ranges from 0 to 100 points. Interpretation of the results: from 90-100 points is an excellent result, 80-90 points is a good result, 60-80 points is a satisfactory result, and below 60 points is a bad result.
PRWE | 3 months after surgery.
  The Patient-Rated Wrist Evaluation (PRWE) score is a highly reliable and valid 15-question questionnaire designed to measure wrist pain and disability in activities of daily living. The PRWE allows patients to assess their own level of pain and disability in the wrist from 0 to 10, and consists of 2 parts: pain and function. The part about pain contains 5 questions, the maximum score in this part is 50, and the minimum is 0. The part about function contains 10 questions divided into 2 parts, i.e. specific activities (6 questions) and usual activities (4 questions). The maximum score in this part is 50, and the minimum is 0.
PRWE | 6 months after surgery.
  The Patient-Rated Wrist Evaluation (PRWE) score is a highly reliable and valid 15-question questionnaire designed to measure wrist pain and disability in activities of daily living. The PRWE allows patients to assess their own level of pain and disability in the wrist from 0 to 10, and consists of 2 parts: pain and function. The part about pain contains 5 questions, the maximum score in this part is 50, and the minimum is 0. The part about function contains 10 questions divided into 2 parts, i.e. specific activities (6 questions) and usual activities (4 questions). The maximum score in this part is 50, and the minimum is 0.

REFERENCES:
- [Background] Court-Brown CM, Caesar B. Epidemiology of adult fractures: A review. Injury. 2006 Aug;37(8):691-7. doi: 10.1016/j.injury.2006.04.130. Epub 2006 Jun 30. PMID 16814787
- [Background] Rundgren J, Bojan A, Mellstrand Navarro C, Enocson A. Epidemiology, classification, treatment and mortality of distal radius fractures in adults: an observational study of 23,394 fractures from the national Swedish fracture register. BMC Musculoskelet Disord. 2020 Feb 8;21(1):88. doi: 10.1186/s12891-020-3097-8. PMID 32035488
- [Background] Ochen Y, Peek J, van der Velde D, Beeres FJP, van Heijl M, Groenwold RHH, Houwert RM, Heng M. Operative vs Nonoperative Treatment of Distal Radius Fractures in Adults: A Systematic Review and Meta-analysis. JAMA Netw Open. 2020 Apr 1;3(4):e203497. doi: 10.1001/jamanetworkopen.2020.3497. PMID 32324239
- [Background] Song J, Yu AX, Li ZH. Comparison of conservative and operative treatment for distal radius fracture: a meta-analysis of randomized controlled trials. Int J Clin Exp Med. 2015 Oct 15;8(10):17023-35. eCollection 2015. PMID 26770293
- [Background] Ju JH, Jin GZ, Li GX, Hu HY, Hou RX. Comparison of treatment outcomes between nonsurgical and surgical treatment of distal radius fracture in elderly: a systematic review and meta-analysis. Langenbecks Arch Surg. 2015 Oct;400(7):767-79. doi: 10.1007/s00423-015-1324-9. Epub 2015 Aug 30. PMID 26318178
- [Background] Chen Y, Chen X, Li Z, Yan H, Zhou F, Gao W. Safety and Efficacy of Operative Versus Nonsurgical Management of Distal Radius Fractures in Elderly Patients: A Systematic Review and Meta-analysis. J Hand Surg Am. 2016 Mar;41(3):404-13. doi: 10.1016/j.jhsa.2015.12.008. Epub 2016 Jan 20. PMID 26810824
- [Background] Armstrong KA, von Schroeder HP, Baxter NN, Zhong T, Huang A, McCabe SJ. Stable rates of operative treatment of distal radius fractures in Ontario, Canada: a population-based retrospective cohort study (2004-2013). Can J Surg. 2019 Dec 1;62(6):386-392. doi: 10.1503/cjs.016218. PMID 31782295
- [Background] Mauck BM, Swigler CW. Evidence-Based Review of Distal Radius Fractures. Orthop Clin North Am. 2018 Apr;49(2):211-222. doi: 10.1016/j.ocl.2017.12.001. PMID 29499822
- [Background] Cazzola M, Bergamaschi G, Melazzini M, Ponchio L, Rosti V, Molinari E. Chronic myelogenous leukemia following radiotherapy and chemotherapy for non-Hodgkin lymphoma. Haematologica. 1990 Sep-Oct;75(5):477-9. PMID 2097266
- [Background] Baron JA, Karagas M, Barrett J, Kniffin W, Malenka D, Mayor M, Keller RB. Basic epidemiology of fractures of the upper and lower limb among Americans over 65 years of age. Epidemiology. 1996 Nov;7(6):612-8. doi: 10.1097/00001648-199611000-00008. PMID 8899387
- [Background] Brogren E, Petranek M, Atroshi I. Incidence and characteristics of distal radius fractures in a southern Swedish region. BMC Musculoskelet Disord. 2007 May 31;8:48. doi: 10.1186/1471-2474-8-48. PMID 17540030
- [Background] Mellstrand-Navarro C, Pettersson HJ, Tornqvist H, Ponzer S. The operative treatment of fractures of the distal radius is increasing: results from a nationwide Swedish study. Bone Joint J. 2014 Jul;96-B(7):963-9. doi: 10.1302/0301-620X.96B7.33149. PMID 24986952
- [Background] Stirling ERB, Johnson NA, Dias JJ. Epidemiology of distal radius fractures in a geographically defined adult population. J Hand Surg Eur Vol. 2018 Nov;43(9):974-982. doi: 10.1177/1753193418786378. Epub 2018 Jul 17. PMID 30016904
- [Background] Solvang HW, Nordheggen RA, Clementsen S, Hammer OL, Randsborg PH. Epidemiology of distal radius fracture in Akershus, Norway, in 2010-2011. J Orthop Surg Res. 2018 Aug 13;13(1):199. doi: 10.1186/s13018-018-0904-0. PMID 30103788
- [Background] Whipple TL. The role of arthroscopy in the treatment of intra-articular wrist fractures. Hand Clin. 1995 Feb;11(1):13-8. PMID 7751326
- [Background] Lutsky K, Boyer MI, Steffen JA, Goldfarb CA. Arthroscopic assessment of intra-articular distal radius fractures after open reduction and internal fixation from a volar approach. J Hand Surg Am. 2008 Apr;33(4):476-84. doi: 10.1016/j.jhsa.2007.12.009. PMID 18406950
- [Background] Jotanović Z, Mamula M, Vlahović T, i sur. Wrist arthroscopy. Medicina Flum 2013;49(3):292- 300.
- [Background] Burnier M, Le Chatelier Riquier M, Herzberg G. Treatment of intra-articular fracture of distal radius fractures with fluoroscopic only or combined with arthroscopic control: A prospective tomodensitometric comparative study of 40 patients. Orthop Traumatol Surg Res. 2018 Feb;104(1):89-93. doi: 10.1016/j.otsr.2017.08.021. Epub 2017 Dec 11. PMID 29241818
- [Background] Geissler WB, Freeland AE, Savoie FH, McIntyre LW, Whipple TL. Intracarpal soft-tissue lesions associated with an intra-articular fracture of the distal end of the radius. J Bone Joint Surg Am. 1996 Mar;78(3):357-65. doi: 10.2106/00004623-199603000-00006. PMID 8613442
- [Background] Ogawa T, Tanaka T, Yanai T, Kumagai H, Ochiai N. Analysis of soft tissue injuries associated with distal radius fractures. BMC Sports Sci Med Rehabil. 2013 Sep 2;5(1):19. doi: 10.1186/2052-1847-5-19. PMID 24004506
- [Background] Swart E, Tang P. The Effect of Ligament Injuries on Outcomes of Operatively Treated Distal Radius Fractures. Am J Orthop (Belle Mead NJ). 2017 Jan/Feb;46(1):E41-E46. PMID 28235122
- [Background] Smeraglia F, Del Buono A, Maffulli N. Wrist arthroscopy in the management of articular distal radius fractures. Br Med Bull. 2016 Sep;119(1):157-65. doi: 10.1093/bmb/ldw032. Epub 2016 Aug 22. PMID 27554281
- [Background] Saab M, Guerre E, Chantelot C, Clavert P, Ehlinger M, Bauer T; SoFCOT. Contribution of arthroscopy to the management of intra-articular distal radius fractures: Knowledge update based on a systematic 10-year literature review. Orthop Traumatol Surg Res. 2019 Dec;105(8):1617-1625. doi: 10.1016/j.otsr.2019.06.016. Epub 2019 Sep 13. PMID 31526708
- [Background] Yamazaki H, Uchiyama S, Komatsu M, Hashimoto S, Kobayashi Y, Sakurai T, Kato H. Arthroscopic assistance does not improve the functional or radiographic outcome of unstable intra-articular distal radial fractures treated with a volar locking plate: a randomised controlled trial. Bone Joint J. 2015 Jul;97-B(7):957-62. doi: 10.1302/0301-620X.97B7.35354. PMID 26130352
- [Background] Kasapinova K, Kamiloski V. Influence of associated lesions of the intrinsic ligaments on distal radius fractures outcome. Arch Orthop Trauma Surg. 2015 Jun;135(6):831-8. doi: 10.1007/s00402-015-2203-0. Epub 2015 Mar 25. PMID 25804372
- [Background] Varitimidis SE, Basdekis GK, Dailiana ZH, Hantes ME, Bargiotas K, Malizos K. Treatment of intra-articular fractures of the distal radius: fluoroscopic or arthroscopic reduction? J Bone Joint Surg Br. 2008 Jun;90(6):778-85. doi: 10.1302/0301-620X.90B6.19809. PMID 18539672
- [Background] Boateng GO, Neilands TB, Frongillo EA, Melgar-Quinonez HR, Young SL. Best Practices for Developing and Validating Scales for Health, Social, and Behavioral Research: A Primer. Front Public Health. 2018 Jun 11;6:149. doi: 10.3389/fpubh.2018.00149. eCollection 2018. PMID 29942800
- [Background] Meinberg EG, Agel J, Roberts CS, Karam MD, Kellam JF. Fracture and Dislocation Classification Compendium-2018. J Orthop Trauma. 2018 Jan;32 Suppl 1:S1-S170. doi: 10.1097/BOT.0000000000001063. No abstract available. PMID 29256945
- [Background] Tsang S, Royse CF, Terkawi AS. Guidelines for developing, translating, and validating a questionnaire in perioperative and pain medicine. Saudi J Anaesth. 2017 May;11(Suppl 1):S80-S89. doi: 10.4103/sja.SJA_203_17. PMID 28616007
- [Background] Sousa VD, Rojjanasrirat W. Translation, adaptation and validation of instruments or scales for use in cross-cultural health care research: a clear and user-friendly guideline. J Eval Clin Pract. 2011 Apr;17(2):268-74. doi: 10.1111/j.1365-2753.2010.01434.x. Epub 2010 Sep 28. PMID 20874835
- [Background] Palmer AK. Triangular fibrocartilage complex lesions: a classification. J Hand Surg Am. 1989 Jul;14(4):594-606. doi: 10.1016/0363-5023(89)90174-3. PMID 2666492
- [Background] Viegas SF, Patterson RM, Peterson PD, Pogue DJ, Jenkins DK, Sweo TD, Hokanson JA. Ulnar-sided perilunate instability: an anatomic and biomechanic study. J Hand Surg Am. 1990 Mar;15(2):268-78. doi: 10.1016/0363-5023(90)90107-3. PMID 2324456
- [Background] Robert H, Lambotte JC, Flicoteaux R. Arthroscopic Measurement of Cartilage Lesions of the Knee Condyle: Principles and Experimental Validation of a New Method. Cartilage. 2011 Jul;2(3):237-45. doi: 10.1177/1947603510388028. PMID 26069582